CLINICAL TRIAL: NCT02274792
Title: A Single-arm Study to Assess the Immunogenicity and Safety of Etanercept Produced Using a Modified Process in Subjects With Plaque Psoriasis
Brief Title: Study to Assess the Immunogenicity and Safety of Etanercept Produced Using a Modified Process in Patients With Plaque Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20101177
Record Dates: First submitted 2014-10-22; First posted 2014-10-24 (Estimated); Results first posted 2016-12-29 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-10

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Etanercept (Experimental): Participants received etanercept 50 mg subcutaneously twice a week (BIW) for 12 weeks followed by 50 mg once a week for an additional 12 weeks.
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — Etanercept produced using the serum free process (SFP)2 was supplied in a single-use 1 mL prefilled syringe for subcutaneous injection.
  Other Names: Enbrel®

SUMMARY:
The purpose of this study is to learn more about the immune response to etanercept produced using a modified process in patients with plaque psoriasis.

DETAILED DESCRIPTION:
This is a multicenter, open-label, single-arm phase 4 study in patients with plaque psoriasis who are etanercept-naïve and who are not receiving methotrexate therapy. The study will consist of a screening period of up to 30 days, a 24-week treatment period and a 30-day follow-up period for safety. Etanercept dosing will follow the recommended label dosing for patients with plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years of age at time of screening.
* Subject is a candidate for systemic therapy or phototherapy in the opinion of the investigator.
* Subject has involved body surface area (BSA) ≥ 10%, static physician global assessment (sPGA) ≥ 3, and Psoriasis Area and Severity Index (PASI) ≥ 10 at screening and at baseline.
* Subject is naïve to etanercept.
* Subject is a candidate for treatment with etanercept in the opinion of the investigator in addition to the caring physician's intent to initiate treatment with etanercept, as applicable.
* Subject is able to self-inject etanercept or have a designee who can do so.
* Subject has not used methotrexate within 4-weeks from the first dose of etanercept.
* Subject has a negative test for hepatitis B surface antigen, hepatitis B core antibody and hepatitis C antibody.
* Subject has no known history of active tuberculosis.
* Subject has a negative test for tuberculosis during screening
* Subject, if female and not at least 2 years postmenopausal or history of hysterectomy, bilateral salpingectomy, or bilateral oophorectomy, has a negative serum pregnancy test ≤ 4 weeks from starting etanercept and a negative urine pregnancy test at baseline (day 1).

Exclusion Criteria:

* Subject has active erythrodermic, pustular, guttate psoriasis, or medication induced psoriasis, or other skin conditions at the time of the screening visit (e.g., eczema) that would interfere with evaluations of the effect of investigational product on psoriasis.
* Subject has any uncontrolled, clinically significant systemic disease (e.g., renal failure, heart failure, hypertension, pulmonary or liver disease, diabetes, anemia).
* Myocardial infarction or unstable angina pectoris within the last year.
* Major chronic inflammatory disease or connective tissue disease other than psoriasis and/or psoriatic arthritis.
* Multiple sclerosis or any other demyelinating disease.
* Active malignancy, including evidence of cutaneous basal or squamous cell carcinoma or melanoma, Merkel cell carcinoma, or history of cancer (other than fully resected and surgically cured cutaneous basal cell and squamous cell carcinoma) within 5 years before the first dose of etanercept. If malignancy occurred more than 5 years ago, documentation of disease-free state since treatment is required.
* Known history of alcoholic hepatitis or immunodeficiency syndromes including human Immunodeficiency virus (HIV) infection.
* Subject has any active infection (including chronic or localized infections) for which anti-infectives were indicated within 4 weeks prior to first dose of etanercept.
* Subject has a serious infection, defined as requiring hospitalization or intravenous (IV) anti-infectives within 8 weeks prior to first dose of etanercept.
* Any condition that, in the opinion of the investigator, might cause this study to be detrimental to the subject.
* Subject has any condition that could, in the opinion of the investigator, compromise the subject's ability to give written consent and/or comply with the study procedures, such as a history of substance abuse or a psychiatric condition.

Ages: 18 Years to 125 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2015-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (40):
- United States (29):
  - Research Site, Mobile, Alabama
  - Research Site, Bakersfield, California
  - Research Site, Beverly Hills, California
  - Research Site, Fremont, California
  - Research Site, Los Angeles, California
  - Research Site, Denver, Colorado
  - Research Site, Aventura, Florida
  - Research Site, Miami, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Carmel, Indiana
  - Research Site, Indianapolis, Indiana
  - Research Site, New Albany, Indiana
  - Research Site, Overland Park, Kansas
  - Research Site, Louisville, Kentucky
  - Research Site, Owensboro, Kentucky
  - Research Site, Rockville, Maryland
  - Research Site, Andover, Massachusetts
  - Research Site, Worcester, Massachusetts
  - Research Site, Clarkston, Michigan
  - Research Site, Omaha, Nebraska
  - Research Site, Verona, New Jersey
  - Research Site, Raleigh, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Johnston, Rhode Island
  - Research Site, Nashville, Tennessee
  - Research Site, Bellaire, Texas
  - Research Site, Dallas, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Norfolk, Virginia
- Canada (11):
  - Research Site, Surrey, British Columbia
  - Research Site, Bathurst, New Brunswick
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Barrie, Ontario
  - Research Site, Courtice, Ontario
  - Research Site, Greater Sudbury, Ontario
  - Research Site, Kingston, Ontario
  - Research Site, Markham, Ontario
  - Research Site, Oakville, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Waterloo, Ontario

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 39 centers in North America (United States and Canada). The first participant enrolled on 29 January 2015 and the last participant was enrolled on 08 May 2015.
Period: Overall Study
Arm/Group | Etanercept
Started | 132
Received Treatment | 131
Completed | 107
Not Completed | 25
Not completed — Withdrawal by Subject | 13
Not completed — Lost to Follow-up | 8
Not completed — Protocol Specified Criteria | 2
Not completed — Sponsor Decision | 2

BASELINE CHARACTERISTICS:
Population: Safety analysis set (all enrolled participants who received ≥ 1 dose of investigational product during the study)
Arm/Group | Etanercept
Number analyzed (Participants) | 131
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (13.2)
Age, Customized [Number; unit: participants]
  < 65 years | 114
  ≥ 65 years | 17
Gender [Count of Participants; unit: Participants]
  Female | 42
  Male | 89
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 8
  Black | 7
  Native Hawaiian or Other Pacific Islander | 1
  White | 112
  Other | 3
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic/Latino | 20
  Not Hispanic/Latino | 111
Duration of Psoriasis [Mean (Standard Deviation); unit: years] | 18.1 (12.6)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Positive Anti-etanercept Binding Antibody Response During the Study
Description: Seroreactivity to etanercept was evaluated using a validated enzyme-linked immunosorbent assay (ELISA).
Time Frame: Blood samples were collected for anti-etanercept antibody analysis before the administration of etanercept at baseline (day 1) and at week 12 and week 24.
Population: Primary Antibody Analysis Set included all enrolled participants who received ≥ 1 dose of investigational product and had both a baseline and ≥ 1 post-baseline serum obtained for anti-etanercept antibody assessment, excluding participants with a negative antibody response at week 12 and missing antibody assessment at week 24.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 106
percentage of participants | 3.8 [1.04 to 9.38]

2. Secondary Outcome: Percentage of Participants With Positive Anti-etanercept Binding Antibody Response at Week 24
Time Frame: Week 24
Population: Participants with available antibody response data at week 24
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 105
percentage of participants | 1.0 [0.02 to 5.19]

3. Secondary Outcome: Percentage of Participants With Positive Anti-etanercept Binding Antibody Response at Week 12
Time Frame: Week 12
Population: Participants with available antibody response data at week 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 120
percentage of participants | 2.5 [0.52 to 7.13]

4. Secondary Outcome: Percentage of Participants With Positive Anti-etanercept Neutralizing Antibody Response at Week 24
Description: Samples confirmed to be positive on the binding assay were subsequently tested in a non-cell based assay to determine neutralizing activity against etanercept.
Time Frame: Week 24
Population: Participants with a positive anti-etanercept antibody binding response at week 24
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 1
percentage of participants | 0.0 [0.00 to 97.50]

5. Secondary Outcome: Percentage of Participants With Positive Anti-etanercept Neutralizing Antibody Response at Week 12
Description: as for outcome 4
Time Frame: Week 12
Population: Participants with a positive anti-etanercept antibody binding response at week 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 3
percentage of participants | 0.0 [0.00 to 70.76]

ADVERSE EVENTS:
Time Frame: From the first dose of investigational product through 30 days after last dose; 28 weeks.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Etanercept
Serious Adverse Events (participants affected / at risk) | 5/131
Other Adverse Events (participants affected / at risk) | 24/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=131)
Myocardial infarction (Cardiac disorders) | 1
Abdominal wall infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=131)
Injection site reaction (General disorders) | 10
Headache (Nervous system disorders) | 7
Psoriasis (Skin and subcutaneous tissue disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.